CLINICAL TRIAL: NCT04611724
Title: A Multicenter Prospective Phase II Study of Modified FOLFIRINOX for 1st Line Treatment for Advanced Urachus Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Green Cross Corporation (Industry); Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jae-Lyun Lee, professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULTIMA
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Urachal Cancer
Keywords: Urachal Cancer; FOLFIRINOX
MeSH Terms: conditions — Urachal cancer | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- FOLFIRINOX (Experimental): oxaliplatin 85 mg/m2 IV over 2 hours leucovorin 400 mg/m2 over 2 hours irinotecan 150 mg/m2 over 90 min, 5-FU continuous infusion 2400 mg/m2 continuous infusion over 46 hours
  Interventions: Drug: FOLFIRINOX

INTERVENTIONS:
Drug: FOLFIRINOX — oxaliplatin 85 mg/m2 IV over 2 hours leucovorin 400 mg/m2 over 2 hours irinotecan 150 mg/m2 over 90 min, 5-FU continuous infusion 2400 mg/m2 continuous infusion over 46 hours

SUMMARY:
This study aims to assess objective response rate of modified FOLFIRINOX in advanced urachaus cancer.

Patients with locally advanced, recurrent, or metastatic urachal carcinoma of bladder, urachal will be enrolled this study.

Modified version of FOLFIRINOX(Oxaliplatin 85 mg/m 2, Leucovorin 400mg/m2 , irinotecan 150mg/m2 and 5-FU 2400mg/m2) with prophylactic pegateograstim will be continued till progression, unacceptable toxicity, or till 12 cycles (24 weeks). Study drugs can be administered after 12 cycles to the subjects with benefit from study medication.

Response evaluation will be done every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of bladder/urachal remnant that is clinically consistent with urachal cancer.

Origin in the anterior wall or dome of the bladder Predominant invasion of muscularis or deeper tissues No obvious origin from the overlying urothelium (relative normal-looking urothelial mucosa) No primary adenocarcinoma elsewhere

* Patients with locally advanced, recurrent, or metastatic disease not amenable to surgery, radiotherapy, or combined modality therapy with curative intent
* No prior systemic therapy for advanced urachal cancer. For recurrent disease, previous 5-FU, oxaliplatin, or irinotecan chemotherapy as neoadjuvant and/or adjuvant aim is allowed if it ended more than 6 months before enrollment.
* Measurable disease according to RECIST v1.1 criteria
* ECOG performance status 0 or 1
* Age 19 years or older
* Adequate cardiac function
* Adequate bone marrow, hepatic, and renal function Hematology
* Life expectancy more than 3 months
* Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Age > 65
* Previous radiotherapy to the only measurable lesion: but previous radiotherapy will be permitted unless the lesion is the only measurable lesion
* Uncontrolled CNS metastasis (brain and/or leptomeningeal metastasis)
* Grade 2 or more peripheral neuropathy
* Diagnosis of any serious secondary malignancy within the last 2 years, except for adequately treated basal cell or squamous cell carcinoma of skin, or in situ carcinoma of cervix uteri or prostate cancer and curatively treated thyroid cancer of any stage.
* Pregnancy or breast feeding, or intention of becoming pregnant during study treatment or within 6 months after final dose
* Other severe acute or chronic medical or psychiatric condition
* Chronic diarrhea
* Clinically significant cardiac disease (heart failure, coronary artery disease, and/or arrhythmia)
* Hypersensitivity to study medication
* treatment with a prohibited medication or anticipation of need for prohibited medication ( section 5.5 )

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 2 years
  Objective response rate

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | every 2 weeks up to 30 weeks.
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Progression-free survival (PFS) | up to 2years.
  Progression-free survival (PFS)
Overall survival (OS), | up to 5 years.
  Overall survival (OS),
Incidence of febrile neutropenia | After study completion (an average of 2 year)
  Incidence of febrile neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: Jae -Lyun Lee, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozaka M, Ishii H, Sato T, Ueno M, Ikeda M, Uesugi K, Sata N, Miyashita K, Mizuno N, Tsuji K, Okusaka T, Furuse J. A phase II study of modified FOLFIRINOX for chemotherapy-naive patients with metastatic pancreatic cancer. Cancer Chemother Pharmacol. 2018 Jun;81(6):1017-1023. doi: 10.1007/s00280-018-3577-9. Epub 2018 Apr 9. PMID 29633005
- [Background] Kume H, Tomita K, Takahashi S, Fukutani K. Irinotecan as a new agent for urachal cancer. Urol Int. 2006;76(3):281-2. doi: 10.1159/000091635. PMID 16601395
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29672836/